CLINICAL TRIAL: NCT07274384
Title: Hyperprogression Upon Cemiplimab Alone or With Chemotherapy in PD-L1 ≥ 50% NSCLC: a Biomarker Guided Phase 2 Trial - HYPERBOLIC Trial
Brief Title: Hyperprogression in PD-L1 ≥ 50% NSCLC: a Biomarker Guided Phase 2 Trial
Acronym: HYPERBOLIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Principal Investigator, Roberto Ferrara, Principal Investigator, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-521583-35-00
Record Dates: First submitted 2025-09-17; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Hyperprogression
Keywords: lung; cancer; hyperprogression; chemotherapy; immunotherapy; carboplatin; cisplatin; pemetrexed; paclitaxel; cemiplimab; risk; immune-checkpoint inhibitors; ldns; CD10-; nsclc; PD-L1; randomized; open-label; Lung Immune Prognostic Index; recist; progression; monotherapy; hpd; non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Disease Progression | interventions — Drug Therapy; cemiplimab; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Intervention Model Description: randomized, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-agent immune-checkpoint inhibitors (Active Comparator): single-agent immune-checkpoint inhibitors (SA-ICI) (Cemiplimab)
  Interventions: Drug: Cemiplimab
- PCT regimens + immune-checkpoint inhibitors (Experimental): PCT regimens will include both carboplatin or cisplatin plus pemetrexed (for non-squamous histology) or paclitaxel (for squamous histology) in combination with cemiplimab
  Interventions: Combination Product: chemotherapy plus cemiplimab

INTERVENTIONS:
Combination Product: chemotherapy plus cemiplimab — Combination of platinum-based chemotherapy (PCT) with ICI. PCT regimens will include both carboplatin or cisplatin plus pemetrexed (for non-squamous histology) or paclitaxel (for squamous histology) in combination with cemiplimab. PCT will be administered for three cycles.
  Other Names: cemiplimab; carboplatin; cisplatin; pemetrexed; paclitaxel
  Arms: PCT regimens + immune-checkpoint inhibitors
Drug: Cemiplimab — single-agent immune-checkpoint inhibitors
  Other Names: libtayo
  Arms: single-agent immune-checkpoint inhibitors

SUMMARY:
In metastatic NSCLC patients with PD-L1 expression ≥50%, a circulating immature (CD10-) LDNs level of ≥30.5% confers a high risk of hyperprogression (HPD) with first line single-agent immune-checkpoint inhibitors (SA-ICI). HPD is defined as a tumor growth rate (TGR) delta ≥50% between pre-treatment and post-treatment, and/or a TGR ratio ≥2. The combination of platinum-based chemotherapy (PCT) with ICI in this setting could prevent the occurrence of HPD and ultimately improve survival outcomes.

This randomized, multicentric, open-label, phase 2 trial will include patients with stage IV NSCL, without targetable oncogene drivers, PD-L1 TPS≥50%, and measurable disease on two CT scans performed before randomization. Participants will be randomized 1:1 to SA-ICI or ICI+PCT. Radiological evaluation will be performed by CT-scan at 6-8 weeks and subsequently according to the local investigators' schedule.

In the SA-ICI arm, ICI regimen will include cemiplimab. In the PCT+ICI arm, PCT regimens will include both carboplatin or cisplatin + pemetrexed (for non-squamous histology) or paclitaxel (for squamous histology) in combination with cemiplimab.

PCT will be administered for three cycles. In case of stable disease or partial response according to RECIST v.1.1, cemiplimab will be performed as monotherapy from the third cycle until disease progression or unacceptable toxicity. If progression according to RECIST v.1.1 or HPD after three cycles of PCT+ICI, patients will be treated with standard second line therapy as local standard of care.

DETAILED DESCRIPTION:
Intervention: PCT plus cemiplimab for 3 cycles followed by cemiplimab in case of absence of PD/HPD. PCT regimens will include both carboplatin (area under the concentration-time curve, 5 mg per milliliter per minute) or cisplatin (75 mg per square meter of body surface area) plus pemetrexed (500 mg per square meter) for non-squamous histology or paclitaxel (200 mg per square meter) for squamous histology. All drugs in the PCT regimens will be administered intravenously every 3 weeks. Cemiplimab 350 mg "flat dose" will be administered intravenously every 3 weeks. Treatment will continue for a maximum of 108 weeks or until progression or unacceptable toxicity.

Comparator: Single-agent cemiplimab. Cemiplimab 350 mg "flat dose" will be administered intravenously every 3 weeks for 108 weeks or until progression or unacceptable toxicity.

Efficacy criteria: The rate of patients experienced HPD or ED will be calculated for both treatment arms.1 HPD is defined as a delta of tumor growth rate (TGR) ≥50% and/or a TGR ratio ≥2. TGR will be computed using RECIST v.1.1 on three consecutive, centrally revised, CT scans (two CT scans before treatment start and one after 7 week ± 5 days from treatment start).

Central review of CT scans will be performed before treatment start and after the first radiological evaluation (before third cycle). RECIST response after the second cycles will be decided according to central review.

ED is defined as tumor-related death within 12 weeks from ICI initiation, in absence of a radiological evaluation performed during ICI.

HPD rate according to definitions proposed by Lo Russo et al., Matos et al.et Saâd-Bouzid et al., will be evaluated as a secondary endpoint.

Efficacy parameters: After the first radiological evaluation performed at 7 weeks ± 5 days from treatment start, subjects will be evaluated by CT scans every 12 weeks ± 28 days according to local investigators' schedule.

CT scans are to be performed until disease progression or until the start of new anticancer treatment, withdrawal of consent, or death, whichever occurs first.

Per RECIST 1.1, the partial and complete response should be confirmed by a repeat tumor imaging assessment not less than 4 weeks from the date the response was first documented.

The enrollment period will last 48 months. The approximate duration of the active study assessments for each patient, including the screening phase, will be 3 months (the time required to confirm HPD occurrence or not). The duration of the active portion of the study will be 48 months, followed by and additional 3 months of follow-up, for a total of 51 months. In both arms, patients will receive treatment for a maximum of 108 weeks or until disease progression or unacceptable toxicity occurs. After the active portion of the study is completed, all patients will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative) has provided documented informed consent to participation to the study and data protection consent form.
2. Male or female aged 18 years or older.
3. ECOG Performance Status of 0 - 2.
4. Pathologically (histologically or cytologically) confirmed diagnosis of stage IV NSCLC (TNM 8th edition), who received no prior systemic treatment for recurrent or metastatic NSCLC. Mixed squamous/non-squamous tumors are eligible.
5. PD-L1 TPS ≥ 50% (by local test).
6. Absence of targetable oncogene alterations (EGFR, ALK, ROS1).
7. Circulating CD10- LDNs >30.5% at screening. LDNs will be defined as CD11b+CD15+ cells among live PBMC. Flow cytometry raw data will be centrally analyzed by the coordinating center.
8. Measurable disease (RECIST 1.1) on two CT scans performed before randomization. The following criteria must be fulfilled:

   * Participants must have at least one measurable lesion that has not been previously treated with radiotherapy.
   * Chest and abdomen scans are mandatory
   * Availability of measurable disease scans to be anonymized and sent for central independent confirmation by a radiologist of the coordinating center.
   * A minimum 2-week interval and a maximum 12-week interval will be acceptable between the two pre-treatment CT scans.
   * Availability to perform the baseline scan within a maximum 4-week interval before treatment start.
9. Patient's willingness to undergo blood draws to provide plasma and blood samples for analysis according to study objectives.
10. Adequate organ and marrow function as defined below:

    * Absolute neutrophil count > 1.5 x 109/L (1500/mm3)
    * Platelets ≥100 x 109/L (100 000/mm3)
    * Haemoglobin ≥9.0 g/dL (5.59 mmol/L)
    * Estimated glomerular filtration rate (according to CDK-EPI equation): ≥ 60ml/min/1.73 m2 for patients receiving cisplatin; ≥30 ml/min/1.73 m2 for patients receiving carboplatin.
    * Serum bilirubin ≤1.5 x upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of hemolysis or hepatic pathology) who will be allowed in consultation with their physician.
    * AST and ALT ≤2.5 x ULN.
11. Absence of a known severe hypersensitivity (≥ Grade 3) to any of the study chemotherapy agents and/or cemiplimab and/or to any of their excipients

Exclusion Criteria:

1. Any infection requiring hospitalization or treatment with IV anti-infectives within 2 weeks of first dose of study medication
2. Known uncontrolled infection with HIV, hepatitis B or hepatitis C infection, diagnosis of immunodeficiency, and/or tuberculosis (active or latent). No serological testing is required unless mandated by local health authority.
3. Administration of live or live-attenuated vaccines within 30 days before the baseline LDNs assessment. Administration of killed vaccines is allowed. Receipt of COVID-19 vaccination within 1 week of planned start of study medication or for which the planned COVID-19 vaccinations would not be completed 1 week prior to start of study medication.
4. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), of active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management.
5. Administration of radiotherapy within 7 days prior to the baseline LDNs assessment.
6. Administration of colony-stimulating factors (e.g., G-CSF, GM-CSF) or recombinant erythropoietin within 28 days prior to the baseline LDNs assessment. Primary prophylaxis with G-CSF and pegylated G-CSF is not allowed. Secondary prophylaxis is not recommended and required case-by-case discussion with the coordinator center before G-CSF administration.
7. Ongoing or recent evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments. The following are not exclusionary: vitiligo, childhood asthma that has resolved, endocrinopathies (such as hypothyroidism or type 1 diabetes) that require only hormone replacement, or psoriasis that does not require systemic treatment.
8. Female patients who are pregnant, breast-feeding, male, or female patients of reproductive potential who are not employing an highly effective method of birth control.
9. Any condition that, in the opinion of the investigator, would interfere with the evaluation of the study drug or interpretation of patient safety or study results.
10. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment (Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable).
11. Allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
HPD rate | up to HPD, end of treatment for a maximum of 108 weeks whichever comes first
  HPD rate, defined as the proportion of patients with a delta of TGR ≥50% or a TGR ratio ≥2 at 7 weeks ± 5 days from randomization
ED rate | up to ED, end of treatment for a maximum of 108 weeks whichever comes first
  ED rate: who died without undergoing a scan after treatment initiation.

SECONDARY OUTCOMES:
Overall survival (OS) | up to HPD, ED, end of treatment for a maximum of 108 weeks whichever comes first
  To compare the activity of cemiplimab+PCT relative to cemiplimab alone.
Progression free survival (PFS) | up to HPD, ED, end of treatment for a maximum of 108 weeks whichever comes first
  To compare the activity and efficacy of cemiplimab+PCT relative to cemiplimab alone
Objective response rate (ORR) | up to HPD, ED, end of treatment for a maximum of 108 weeks whichever comes first
  To compare the activity of cemiplimab+PCT relative to cemiplimab alone.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 90 days after the last dose of study treatment
  Summary of adverse events (AE), with a focus on TRAEs coded based upon the Medical Dictionary for Regulatory Activities (MedDRA) and graded based upon CTCAE, ver. 5.0.

OTHER OUTCOMES:
Exploratory baseline and dynamic characterization of patients' tissue and circulating clinical and radiological features correlated with HPD occurrence, according to treatment arm | through study completion, an avarage of 3 years
  To characterize how treatments with cemiplimab alone and cemiplimab+PCT modulate circulating or tissue features of HPD, clinical, radiological, and biological
Exploratory characterization of clinical, radiological, and biological patients' features correlated with HPD occurrence. | through study completion, an avarage of 3 years
  To characterize how treatments with cemiplimab alone and cemiplimab+PCT modulate circulating or tissue features of HPD
HPD rate among patients not meeting inclusion criterion 7 | through study completion, an avarage of 3 years
  To characterize HPD rate among patients not meeting inclusion criterion 7 (circulating CD10- LDNs >30.5% at screening).